CLINICAL TRIAL: NCT07238166
Title: Benign Versus Malignant Causes of Intussuception in Adults : A Prospective Study in Assiut University Hospital
Brief Title: Benign Versus Malignant Causes of Intussuception in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew gamal fikry, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Intussusception in adult
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Intussusception (IS)
Keywords: in adult
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patient with intussusception (Other): Adult patient with intussusception will undergo surgical resection followed byhistopathological evaluation to determine the underlying causes ( benign or malignant )
  Interventions: Procedure: surgical resection and histopathological examination

INTERVENTIONS:
Procedure: surgical resection and histopathological examination — Adult patient diagnosed with intussusception will undergo surgical resection of affected bowel segment under general anathesia . the resected specimens will be sent for histopathological evalution to determine the underlying cause , whether benign (e.g lipoma , polyp )or malignant (e.g adenocarcinama , lymphoma ). operative finding , postoperative outcome , and pathology results will be recorded and analyzed

SUMMARY:
The aim of this study is to evaluate adult intussecption :

* Prevalence of benign vs malignant causes.
* Distribution by anatomical type.
* Clinical presentation patterns.
* Diagnostic accuracy of imaging.
* Surgical approach and outcomes.
* Length of hospital stay, complications, recurrence

DETAILED DESCRIPTION:
Intussusception is a condition characterized by the invagination of one segment of the intestine into another, leading to obstruction and potentially ischemia (1). While intussusception is relatively common in the pediatric population, it is considered a rare clinical entity in adults, accounting for only 1-5% of all cases and approximately 1% of intestinal obstructions in the adult population. The etiology, clinical presentation, and management of adult intussusception differ significantly from pediatric cases, necessitating a distinct clinical approach (2).

In contrast to children, where most cases are idiopathic, adult intussusception is commonly associated with an underlying pathological lead point. In approximately 70-90% of adult cases, a structural lesion can be identified as the cause of the intussusception (3). These lesions may be benign or malignant in nature and understanding the incidence of each is important for appropriate diagnosis and treatment planning (4).

In general, intussusceptions involving the small intestine are more likely to be caused by benign lesions such as lipomas, polyps, or Meckel's diverticulum, whereas those involving the colon have a higher likelihood of being associated with malignancy, especially primary adenocarcinoma (5).

Adult intussusception poses a diagnostic challenge due to its nonspecific and often chronic symptoms, which may include intermittent abdominal pain, nausea, vomiting, gastrointestinal bleeding, or signs of partial bowel obstruction (6).

The advent of advanced imaging techniques, particularly abdominal computed tomography (CT), has improved the preoperative diagnosis of this condition (7). However, surgical exploration remains the definitive diagnostic and therapeutic modality, especially given the high probability of underlying malignancy (8).

Despite advancements in diagnostic imaging and surgical techniques, there remains a lack of general agreement regarding the optimal management of adult intussusception, particularly concerning the necessity and extent of bowel resection when a benign cause is suspected (9). Moreover, data on the relative incidence of benign versus malignant causes vary widely across regions, institutions, and populations.

This study aims to evaluate adult intussecption, prevalence of benign versus malignant causes in AUH.

ELIGIBILITY:
a. Inclusion criteria:

* Age ≥ 19 years.

  • Confirmed diagnosis of intussusception by: Imaging (CT , ultrasound , or barium studies) Intraoperative findings,
  * Patients managed surgically with documented follow-up and final diagnosis. b. Exclusion criteria:
  * Patients with incomplete records or lost to follow-up
* Intussusception diagnosed radiologically but resolved spontaneously without confirmatory intervention or follow-up

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of benign versus malignant causes | 2 weeks after surgical resection
  Histopathological examination of resected bowel specimens will determine whether the cause of intussusception is benign (e.g., lipoma, polyp) or malignant (e.g., adenocarcinoma, lymphoma). The frequency and percentage of each category will be calculated

SECONDARY OUTCOMES:
Correlation between preoperative imaging findings and histopathological results Description | At the time of diagnosis (preoperative period )
  Evaluate the diagnostic accuracy of preoperative imaging (CT scan findings such as target sign, mass lesion) in predicting benign or malignant pathology

OTHER OUTCOMES:
Operative findings | During intraoperative period
  To record intraoperative findings including location of intussusception (small bowel, ileocecal, colocolic), presence of lead point, bowel viability, and type of surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of general surgury Assiut uneversity hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Su T, He L, Zhou T, Wu M, Guo Y, Wang Q, Jiang J, Cao X. Most Adult Intussusceptions are Caused by Tumors: A Single-Centre Analysis. Cancer Manag Res. 2020 Oct 12;12:10011-10015. doi: 10.2147/CMAR.S268921. eCollection 2020. PMID 33116857